CLINICAL TRIAL: NCT01813097
Title: Combination Iodine 125 Seed Implants and LHRH Agonists for Locally Advanced (Stage T3) Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xu Yong, director, Chinese PLA General Hospital
Other Study IDs: D8664C00011
Record Dates: First submitted 2013-03-12; First posted 2013-03-18 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2008-02

CONDITIONS: Prostate Cancer
Keywords: To detective the effect of the treatment of combination iodine 125 seed implants and LHRH agonists for the patients with locally advanced prostate cancer.
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- combination iodine 125 seed implants: 30 cases should be treated with iodine 125 seed implants 0.5 mc transperineal prostate implant +Zoladex 3.6mg im 1/28d (LHRH agonist, 3.6mg subcutaneous injection 1/4weeks).
- LHRH agonists: 30 cases should be treated with Zoladex 3.6mg im 1/28d (LHRH agonist, 3.6mg subcutaneous injection 1/4weeks).

SUMMARY:
Patients with prostate cancer should have the following examination including biopsy, serum PSA volume, prostate CT scan or MRI, bone scan, abdomen ultrasound, chest X ray, blood biochemistry, blood rout, ECG and testosterone.

Two groups:

First group:30 cases should be treated with iodine 125 seed implants 0.5 mc transperineal prostate implant +Zoladex 3.6mg im 1/28d (LHRH agonist, 3.6mg subcutaneous injection 1/4weeks).

Second group: 30 cases should be treated with Zoladex 3.6mg im 1/28d (LHRH agonist, 3.6mg subcutaneous injection 1/4weeks).

PFS and PSA level will be the primary variables.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. T2c-T3b N0 M0 (biopsy、 bone scan、 CT、 MRI)
3. No Metastasis (bone scan、 CT、 MRI)
4. PSA level>10ng/ml
5. Histological or cytological confirmation of prostate cancer
6. Able to understand and comply with the requirements of the study

Exclusion Criteria:

1. Having been treated with external radiation therapy or chemistry therapy.
2. Clinical relevant disease and/or abnormalities (past or present), eg, significant cardiovascular, renal or liver disease, malignancy, gastro-intestinal disorders, or other conditions which could affect the absorption/elimination of drugs.
3. Alanine amino transferase (ALT) or aspartate amino transferase (AST) greater than 2 times the upper limit of normal (ULN) at screening findings that make it undesirable for the patient to participate in the study in the opinion of the investigator(s)
4. In the opinion of the investigator(s), any evidence of severe or uncontrolled systemic disease (eg, currently unstable or unresolved respiratory, cardiac, hepatic, or renal disease).
5. Contra-indications (eg, known or suspected allergy) to GnRH antagonists or excipients(non-active ingredients of investigational product).
6. Treatment with a non-approved or investigational drug within 30 days before study entry.
7. Bibulosity or drug abuse.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subject number: <<60>>
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-02; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To detective the effect of the treatment of combination iodine 125 seed implants and LHRH agonists for the patients with locally advanced prostate cancer. | two years